CLINICAL TRIAL: NCT03414697
Title: Transplantation of Umbilical Cord-derived Mesenchymal Stem Cells Via Different Routes for the Treatment of Cerebral Palsy in Children
Brief Title: Transplantation of Umbilical Cord-derived Mesenchymal Stem Cells Via Different Routes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Liu Jing, Principal Investigator, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FirstHospitalDalianMU004
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy
Keywords: umbilical cord-derived mesenchymal stem cells; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Other): Routine rehabilitation treatments
  Interventions: Other: Control group
- Intravenous UC-MSCs group (Experimental): Injection of UC-MSCs via the peripheral vein.
  Interventions: Procedure: UC-MSCs
- Intrathecal UC-MSCs group (Experimental): Injection of UC-MSCs via the intrathecal route.
  Interventions: Procedure: UC-MSCs
- Intranasal UC-MSCs group (Experimental): Injection of UC-MSCs via the nasal route.
  Interventions: Procedure: UC-MSCs

INTERVENTIONS:
Other: Control group — The control group received routine rehabilitation treatments including acupuncture, massage, Bobath therapy, and Vojat therapy.
  Arms: Control group
Procedure: UC-MSCs — Injection of umbilical cord-derived mesenchymal stem cells (UC-MSCs) (at least 1×10^7), once every 2 weeks, one course of treatment including two injections within 4 weeks, a total of two courses of treatment.
  Arms: Intranasal UC-MSCs group; Intrathecal UC-MSCs group; Intravenous UC-MSCs group

SUMMARY:
To preliminarily evaluate the efficacy and safety of umbilical cord-derived mesenchymal stem cells (UC-MSCs), and compare the efficacy of UC-MSCs administered through the intravenous, intrathecal, and intranasal routes, in the treatment of cerebral palsy in children.

DETAILED DESCRIPTION:
Cerebral palsy refers to a neurological disorder caused by a non-progressive brain injury or malformation that occurs in early childhood. It can result in central motor deficits, developmental retardation, abnormal posture, abnormal muscular strength, abnormal muscle tone and/or dysreflexia. It has a high disability rate. There is currently no effective treatment for cerebral palsy. Conventional treatments for cerebral palsy are often tiresome and expensive and have a slow onset of action. Stem cells have been recently used in the treatment of cerebral palsy. This provides a novel method for the treatment of cerebral palsy. According to the existing clinical studies, neural stem cells, bone marrow-derived mesenchymal stem cells, and umbilical cord-derived mesenchymal stem cells (UC-MSCs) are mainly used as the seed cells for the treatment of cerebral palsy. UC-MSCs are the most promising seed cells for the treatment of cerebral palsy because of the advantages including rich sources, ease of harvesting, short doubling time, low immunogenicity, long-time survival post-transplantation, and no ethical issues. UC-MSCs have been widely used to treat Parkinson's disease, rheumatoid arthritis, traumatic brain injury, aplastic anemia, and decompensated liver disease. However,only two studies, and performed only in China, are reported on the treatment of cerebral palsy with UC-MSCs. One from the Hospital 463 of PLA reported 51 patients with cerebral palsy whose symptoms had not been obviously improved after 1 year of rehabilitative treatment. These patients received intrathecal injection of UC-MSCs for three times, once a week, followed by one injection of UC-MSCs via the peripheral vein in the fourth week. Four UC-MSCs injections, once per week, were considered as one course of treatment. Activities of daily living scale score was compared between before and after treatment to evaluate efficacy. Another study is a case report from China. In this report, a combined intravenous and intrathecal injection of UC-MSCs was used to treat cerebral palsy in a 5-year-old child. 28-month follow-up results revealed that the child's gross motor function, immune function, muscle strength, and language ability improved and adverse reactions were not obvious.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hypoxic/ischemic cerebral palsy, primarily including birth asphyxia and premature children
* Patients with spastic quadriplegia
* Patients with moderate to severe cerebral palsy, GMFM scores of 2-3
* Age at 2-18 years
* Provision of signed informed consent by legal representatives of the child prior to start of the study

Exclusion Criteria:

* Those with systemic diseases that likely interfere with the treatment or child's compliance
* Those complicated by life-threatening diseases of any organ
* Those with brain deformity
* Those with uncontrolled epilepsy
* Those with abnormal behavior or mood disorders
* Those with allergies especially those who are allergic to blood products
* Those are infected with infectious diseases
* Those who had underwent a craniocerebral surgery in other clinical trials

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The Gross Motor Function Measure (GMFM)-88 item score | 12 months after 2 courses of treatment with UC-MSCs.
  a 4-point scale that is divided into five categories including lying and rolling, sitting, crawling and kneeling, standing, walking, running, and jumping. A score of 0 indicates that the child does not initiate the task; 1 indicates that the child initiates the task (completes < 10% of the activity); 2 indicates that the child partially completes the task (completes from 10 to 99% of the activity); 3 indicates that the child completes the task (100%). The sum of score of the five categories is used as the evaluation outcome.It is used to evaluate gross motor function.

SECONDARY OUTCOMES:
Fine Motor Function Measure scale (FMFM) score | 1, 3, 6, 9 and 12 months after 2 courses of treatment with UC-MSCs.
  To evaluate fine motor function.The scale is divided into 45 items covering visual tracing (7 items), upper extremity range of motion (8 items), grab ability (8 items), operational ability (10 items), and hand-eye coordination (12 items). The FMFM is a 4-point scale with the score range of 0-3. The original total score is 135. The summed score for evaluating fine motor function measure is 0-100.
The Modified Ashworth scale (MAS) score | 1, 3, 6, 9 and 12 months after 2 courses of treatment with UC-MSCs.
  To evaluate muscle tone. The MAS score is divided into six grades: 0, 1, 1+, 2, 3 and 4. Passive full ranges of motion exercises are performed by moving the knee and ankle until the patient feel a slight resistance from hamstrings and plantar flexor muscles (soleus muscle and gastrocnemius muscle). The average score is calculated across three repeated measurements.
Gesell Development Schedule score | 1, 3, 6, 9 and 12 months after 2 courses of treatment with UC-MSCs.
  To evaluate neurobehavioral development.
Incidence of adverse reactions | 1, 3, 6, 9 and 12 months after 2 courses of treatment with UC-MSCs.
  Liver and kidney dysfunction, fever, infection, vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, Ph.D, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China